CLINICAL TRIAL: NCT03544437
Title: Prospective Clinical Trial of the Feasibility and Safety of Extraperitoneal Laparoscopic Extended Retroperitoneal Lymph Node Dissection at Time of Nephroureterectomy for Upper Tract Urothelial Carcinoma
Brief Title: Feasibility and Safety of Extraperitoneal Laparoscopic Extended Retroperitoneal Lymph Node Dissection at Time of Nephroureterectomy for Upper Tract Urothelial Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: UTUC-LND collaboration 2
Record Dates: First submitted 2018-05-19; First posted 2018-06-01 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Upper Tract Urothelial Carcinoma
Keywords: lymph node dissection; upper tract urothelial carcinoma; nephroureterectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: extraperitoneal laparoscopic extended retroperitoneal lymph node dissection — All patients underwent extraperitoneal laparoscopic RNU with bladder cuff excision with concomitant extended RPLND performed by one of two urology surgeons at Renji Hospital.
  The anatomical boundaries of the lymph node dissection were deﬁned by the ipsilateral side of UUT-UC. In patients with right-sided UUT-UC, the template of dissection consisted of (i) right perihilar lymph nodes, (ii) paracaval lymph nodes, (iii) interaortocaval lymph nodes and (iv) right pelvic lymph nodes (common, external and obturator lymph nodes).
  In patients with left-sided UUT-UC, the template of dissection included (i) left perihilar lymph nodes, (ii) para-aortic lymph nodes, and (iii) left pelvic lymph nodes (common, external and obturator lymph nodes ). Lymph node specimens were sampled "en bloc" with surrounding adipose tissue, and were sent to pathological examination as individual packets with the surrounding adipose tissue.

SUMMARY:
Extended pelvic lymph node dissection in bladder carcinoma provides staging and, in selected patients, a survival beneﬁt. Recent studies showed the therapeutic beneﬁt of retroperitoneal lymph node dissection (RPLND) in advanced stage of upper tract urothelial carcinoma (UTUC). Also laparoscopic extended RPLND is still a technical challenge in urology, considering the high rate of severe complications and difﬁculties in manipulation. In Renji Hospital, laparoscopic extended RPLND at time of nephroureterectomy was performed via an extraperitoneal approach, avoiding interference with abdominal organs and achieving better exposure.The aim of the present study was to determine the safety and feasibility of performing an extraperitoneal laparoscopic extended RPLND at the time of radical nephroureterectomy (RNU) for UTUC in a prospectively collected cohort of patients.

DETAILED DESCRIPTION:
Similar to urothelial carcinoma of the bladder (UCB), UTUC can follow routes of metastases to involve regional lymph nodes. Nodal metastasis is an adverse prognostic indicator and results in poor outcome, irrespective of the use of systemic chemotherapy or radiation. The ' gold standard ' treatment for UUT-UC is RNU.

Extended pelvic lymph node dissection in bladder carcinoma provides staging and, in selected patients, a survival beneﬁt. Recent studies showed the therapeutic beneﬁt of RPLND in advanced stage urothelial carcinoma of the upper urinary tract, but there is still a lack of prospective studies. Thus, the current guideline recommends lymph node dissection for invasive UCUT on the basis of insufﬁcient evidence. But no prospective studies have standardized the ideal extent of RPLND or the optimum number of total lymph nodes that should be removed in patients with UUT-UC. Also more and more interest has been paid to establish standardized node dissection templates.

Also laparoscopic extended RPLND is still a technical challenge in urology, considering the high rate of severe complications and difﬁculties in manipulation. In Renji Hospital, laparoscopic extended RPLND at time of nephroureterectomy was performed via an extraperitoneal approach, avoiding interference with abdominal organs and achieving better exposure.

The aim of the present study was to determine the safety and feasibility of performing an extraperitoneal laparoscopic extended RPLND at the time of RNU for UTUC in a prospectively collected cohort of patients.

ELIGIBILITY:
Inclusion Criteria:

* clinically diagnosed with upper tract urothelial carcinoma
* have no distant metastasis
* have an ECOG 0 to 2
* expected to receive radical nephroureterectomy

Exclusion Criteria:

* had no previous abdominal surgeries
* contra-indications to laparoscopic surgery (e.g. severe chronic obstructive pulmonary disease)
* patients with cT4 disease before surgery

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients who are clinically diagnosed with upper tract urothelial carcinoma and expected to receive radical nephroureterectomy will be the candidates for this study. They will be informed about this study and told about the pros and cons of extraperitoneal laparoscopic extended RPLND. If they were willing to attend this study, chest CT scan and other imaging method would be used to exclude out the distant metastasis.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-05-21 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
Perioperative complications rate | 90 days
  Perioperative complications were evaluated up to 90 days after surgery, and were graded by Clavien-Dindo classiﬁcation.

SECONDARY OUTCOMES:
Operating time | during surgery
  Operating time
Estimate blood loss | during surgery
  Estimate blood loss during surgery
length of stay | 1 month
  The length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xue, M.D, Principal Investigator — Renji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang J, Qian H, Yuan Y, Cai X, Chen Y, Zhang J, Kong W, Wu X, Cao M, Huang Y, Chen H, Xue W. Prospective Clinical Trial of the Oncologic Outcomes and Safety of Extraperitoneal Laparoscopic Extended Retroperitoneal Lymph Node Dissection at Time of Nephroureterectomy for Upper Tract Urothelial Carcinoma. Front Oncol. 2022 Feb 24;12:791140. doi: 10.3389/fonc.2022.791140. eCollection 2022. PMID 35280720